CLINICAL TRIAL: NCT03593655
Title: A Phase 2a Crossover Trial Evaluating the Safety of and Adherence to a Vaginal Matrix Ring Containing Dapivirine and Oral Emtricitabine/Tenofovir Disoproxil Fumarate in an Adolescent and Young Adult Female Population
Brief Title: Evaluating the Safety of and Adherence to a Vaginal Matrix Ring Containing Dapivirine and Oral Emtricitabine/Tenofovir Disoproxil Fumarate in an Adolescent and Young Adult Female Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MTN-034; 12066 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Results first posted 2023-02-03 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence A: Dapivirine vaginal ring + FTC/TDF (Experimental): Participants will receive one 25 mg dapivirine vaginal ring inserted vaginally each month for 24 weeks, followed by one FTC/TDF oral tablet taken by mouth daily for 24 weeks, followed by participant's choice of either or neither study product for 24 weeks.
  Interventions: Device: Dapivirine vaginal ring; Drug: FTC/TDF
- Sequence B: FTC/TDF + Dapivirine vaginal ring (Experimental): Participants will receive one FTC/TDF oral tablet taken by mouth daily for 24 weeks, followed by one 25 mg dapivirine vaginal ring inserted vaginally each month for 24 weeks, followed by participant's choice of either or neither study product for 24 weeks.
  Interventions: Device: Dapivirine vaginal ring; Drug: FTC/TDF

INTERVENTIONS:
Device: Dapivirine vaginal ring — Vaginal ring containing 25 mg of dapivirine
Drug: FTC/TDF — Tablet containing 200 mg FTC/300 mg TDF
  Other Names: Emtricitabine/Tenofovir Disoproxil Fumarate; Truvada

SUMMARY:
The purpose of this study is to evaluate the safety of and adherence to a vaginal matrix ring (VR) containing dapivirine and oral emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) in adolescent and young adult females.

DETAILED DESCRIPTION:
This study will evaluate the safety of and adherence to a vaginal matrix ring (VR) containing dapivirine and oral emtricitabine/tenofovir disoproxil fumarate (FTC/TDF) in adolescent and young adult females.

The study will enroll healthy, HIV-uninfected adolescent and young adult females between 16 and 21 years of age. Participants will be randomized to one of two sequences of one VR containing 25 mg of dapivirine to be inserted monthly for 24 weeks and one 200 mg FTC/300 mg TDF oral tablet taken daily for 24 weeks. After completing the randomized sequence of two study product use periods, participants will then select between the two study products to use in the final 24 weeks of the trial. Participants will be able to choose either or neither study product during the third product use period. The study includes approximately 76 weeks of follow-up per participant.

Participants will attend monthly study visits, which may include behavioral assessments/counseling; physical and pelvic examinations; and blood, urine, and pelvic sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Age 16 through 21 years (inclusive) at Enrollment, verified per site standard operating procedures (SOPs).
* Able and willing to provide informed consent, and if under the legal age of consent be able to provide informed assent and obtain parental or guardian permission/consent, to be screened for and to enroll in MTN-034 (as specified in site SOP).
* Able and willing to provide adequate locator information, as defined in site SOPs.
* Able and willing to comply with all study procedural requirements.
* Per participant report at Screening, post-menarche.
* HIV-uninfected based on testing performed at Screening and Enrollment (per protocol algorithms found in the study protocol).
* Per participant report at Screening, history of at least one episode of sexual intercourse in participant's lifetime.
* Negative pregnancy test at Screening and Enrollment.
* Per participant report, use of an effective method of contraception for at least two months prior to Enrollment, and intending to continue use of an effective method for the duration of study participation; effective methods include:

  * hormonal methods (except contraceptive ring).
  * intrauterine device (IUD).
  * Note: Participant must be on the same contraception method for at least the two months prior to Enrollment.
* Per participant report at Screening, willing to abstain from inserting anything into the vagina for 72 hours prior to each study visit, including receptive intercourse.

  * Note: In the event the VR has been expelled and requires reinsertion, repositioning the VR is permitted.
  * Note: Participant use of tampons is permitted at any time during the study.
* At Screening and Enrollment, agrees not to participate in other research studies involving drugs, medical devices, vaginal products, or vaccines for the duration of study participation, unless approved by the Protocol Safety Review Team (PSRT).

Exclusion Criteria:

* Per participant report at Screening and Enrollment, intends to do any of the following during the study participation period:

  * become pregnant.
  * access and/or use oral PrEP outside the context of study participation.
  * relocate away from the study site.
  * travel away from the study site for a time period that would interfere with product resupply and study participation.
* At Screening or Enrollment, has a positive HIV test.
* Diagnosed with urinary tract infection (UTI), pelvic inflammatory disease (PID), sexually transmitted infection (STI) or reproductive tract infection (RTI) requiring treatment per World Health Organization (WHO) guidelines at Screening or Enrollment.

  * Note: Otherwise eligible participants diagnosed during screening with a UTI, PID or STI/RTI requiring treatment per WHO guidelines - other than asymptomatic bacterial vaginosis (BV) and asymptomatic candidiasis - are offered treatment consistent with WHO recommendations. If treatment is completed and symptoms have resolved within 70 days of obtaining informed assent/consent for screening, the participant may be enrolled. Genital warts requiring treatment also must be treated prior to enrollment. Genital warts requiring therapy are defined as those that cause undue burden or discomfort to the participant, including bulky size, unacceptable appearance, or physical discomfort.
* At Enrollment, has a clinically apparent Grade 2 or higher pelvic exam finding.

  * Note: Cervical friability bleeding associated with speculum insertion and/or specimen collection judged to be within the range of normal according to the clinical judgment of the Investigator of Record (IoR)/designee is considered expected non-menstrual bleeding and is not exclusionary.
  * Note: Otherwise eligible participants with exclusionary pelvic exam findings may be enrolled/randomized after the findings have improved to a non-exclusionary severity grading or resolved. If improvement to a non-exclusionary grade or resolution is documented within 70 days of providing informed assent/consent for screening, the participant may be enrolled.
* Participant report and/or clinical evidence of any of the following:

  * Known adverse reaction to any of the study products (ever).
  * Known adverse reaction to latex and polyurethane (ever).
  * Symptoms suggestive of acute HIV infection at Screening or Enrollment.
  * Non-therapeutic injection drug use in the 12 months prior to Enrollment.
  * Use of HIV PEP and/or PrEP within the 3 months prior to Enrollment.
  * Currently breastfeeding.
  * Last pregnancy outcome within 8 weeks or less of Enrollment.
  * Participation in any other research study involving drugs, medical devices, vaginal products or vaccines within 60 days of Enrollment.
  * At Enrollment, as determined by the IoR/designee, has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease.
* Has any of the following laboratory abnormalities at Screening Visit:

  * Positive for hepatitis B surface antigen (HBsAG).
  * Hemoglobin Grade 2 or higher.
  * Calculated creatinine clearance less than 60 mL/min by the Schwartz Equation.

    * Note: Otherwise eligible participants with an exclusionary test may be re-tested during the screening process; re-testing procedure details can be found in the MTN-034 Study Specific Procedures (SSP) Manual. If improvement to a non-exclusionary grade or resolution is documented within 70 days of providing informed assent/consent for screening, the participant may be enrolled.
* Has any other condition that, in the opinion of the IoR/designee, would preclude informed assent/consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 247 (Actual)
Dates: Start 2019-01-14 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gonasagrie Nair, MBChB, MPH, Study Chair — Emavundleni Research Centre
Locations (4):
- South Africa (2):
  - Wits Reproductive Health and HIV Institute CRS (WRHI CRS), Johannesburg, Gauteng
  - Emavundleni CRS, Cape Town, Western Cape
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Uganda
- Spilhaus CRS, Southerton, Harare, Zimbabwe

REFERENCES:
- [Derived] Friedland BA, Browne EN, Roberts ST, Ngure K, Nakalega R, Macdonald P, Mpongo CN, Tenza S, Mhlanga N, Szydlo D, Johnson S, McClure T, Nair G, Celum C, Hillier SL, van der Straten A; MTN-034 REACH clinical trial team. Higher Acceptability of the Monthly Dapivirine Ring Versus Daily Oral Pre-Exposure Prophylaxis Among Adolescent Girls and Young Women in Sub-Saharan Africa in the REACH Trial. J Acquir Immune Defic Syndr. 2025 Dec 15;100(5):415-424. doi: 10.1097/QAI.0000000000003756. PMID 40875480
- [Derived] Shapley-Quinn MK, Tenza S, Jensen D, Tauya T, Mampuru L, Etima J, Kemigisha D, Atujuna M, Soto-Torres L, Johnson S, Mpongo N, Mhlanga N, Ngure K, van der Straten A. Adolescent Girls and Young Women Overcoming Adherence Challenges with Vaginal and Oral PrEP Use: A Longitudinal Qualitative Study from a Crossover Trial in South Africa, Uganda, and Zimbabwe. AIDS Behav. 2024 Dec;28(12):4209-4223. doi: 10.1007/s10461-024-04503-y. Epub 2024 Sep 30. PMID 39343865
- [Derived] Nair G, Celum C, Szydlo D, Brown ER, Akello CA, Nakalega R, Macdonald P, Milan G, Palanee-Phillips T, Reddy K, Tahuringana E, Muhlanga F, Nakabiito C, Bekker LG, Siziba B, Hillier SL, Baeten JM, Garcia M, Johnson S, McClure T, Levy L, Livant E, Jacobson C, Soto-Torres L, van der Straten A, Hosek S, Rooney JF, Steytler J, Bunge K, Parikh U, Hendrix C, Anderson P, Ngure K; REACH Protocol Team. Adherence, safety, and choice of the monthly dapivirine vaginal ring or oral emtricitabine plus tenofovir disoproxil fumarate for HIV pre-exposure prophylaxis among African adolescent girls and young women: a randomised, open-label, crossover trial. Lancet HIV. 2023 Dec;10(12):e779-e789. doi: 10.1016/S2352-3018(23)00227-8. Epub 2023 Oct 25. PMID 37898146
- [Derived] Young AM, Mancuso N, Atujuna M, Tenza S, Chitukuta M, Kemigisha D, Ngure K, van der Straten A, Garcia M, Szydlo D, Soto-Torres L, Roberts ST. Adolescent Girls and Young Women's Experiences with Disclosing Oral PrEP or Dapivirine Vaginal Ring Use: a Multi-Country Qualitative Analysis. AIDS Behav. 2023 Dec;27(12):3941-3951. doi: 10.1007/s10461-023-04109-w. Epub 2023 Jul 1. PMID 37392268

RESULTS

PARTICIPANT FLOW:
Period: First Product Use Period
Arm/Group | Sequence A: Dapivirine Vaginal Ring + FTC/TDF | Sequence B: FTC/TDF + Dapivirine Vaginal Ring
Started | 124 | 123
Completed | 122 | 119
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 3
Period: Second Product Use Period
Arm/Group | Sequence A: Dapivirine Vaginal Ring + FTC/TDF | Sequence B: FTC/TDF + Dapivirine Vaginal Ring
Started | 122 | 119
Completed | 120 | 118
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Period: Third Product Use Period
Arm/Group | Sequence A: Dapivirine Vaginal Ring + FTC/TDF | Sequence B: FTC/TDF + Dapivirine Vaginal Ring
Started | 120 | 118
Always Chose Dapivirine Vaginal Ring | 66 | 71
Always Chose FTC/TDF | 35 | 27
At Least One Switch (This category includes participants who switched between the ring and FTC/TDF, as well as participants who switched between using one/both of the products and using neither product.) | 17 | 13
Never Chose Either Product | 2 | 7
Completed | 119 | 114
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence A: Dapivirine Vaginal Ring + FTC/TDF | Sequence B: FTC/TDF + Dapivirine Vaginal Ring | Total
Number analyzed (Participants) | 124 | 123 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.3 (1.4) | 18.2 (1.4) | 18.3 (1.4)
Age, Customized [Count of Participants; unit: Participants]
  16-17 years | 41 | 44 | 85
  18-19 years | 57 | 57 | 114
  20-21 years | 26 | 22 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 123 | 247
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 124 | 123 | 247
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 120 | 119 | 239
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Uganda | 30 | 30 | 60
  Zimbabwe | 30 | 30 | 60
  South Africa | 64 | 63 | 127

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 or Higher Adverse Events (AEs)
Description: During participants' first year on study (i.e., during first and second product use periods) participants were randomized to use either the dapivirine vaginal ring for 6 months followed by FTC/TDF for 6 months or vice versa. All AEs were reported as per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events. AEs that were graded as at least Grade 2 (i.e., "moderate" or higher) were classified into the two periods based on reported date of AE onset, with AEs occurring between the participant's randomization date and the date 30 days after their Week 24 visit classified into Period 1, and AEs occurring between their Week 24 visit and the date 30 days after their Week 48 visit classified into Period 2. AEs occurring within 30 days of the Week 24 visit were counted in both periods.
  This is the number of participant-periods with at least one grade 2 or higher AE by product (combining the two product use periods).
Time Frame: Study periods 1 and 2
Population: All participants who attended at least one visit during the product use period where they were randomized to receive the product (e.g., a participant randomized to Sequence A would be in the analysis population for dapivirine vaginal ring due to being randomized, and would be in the analysis population for FTC/TDF if they attended any study visits during the second product use period).
Measure: Count of Participants; unit: Participants
Groups:
- Dapivirine Vaginal Ring: The period during the first two product use periods where the participant was randomized to use the dapivirine ring. This is the first product use period for participants randomized to Sequence A (i.e., participants who were randomized to receive the dapivirine vaginal ring during their first product use period) or the second product use period for participants randomized to Sequence B (i.e., participants who were randomized to receive the dapivirine vaginal ring during their second product use period).
- FTC/TDF: The period during the first two product use periods where the participant was randomized to use FTC/TDF. This is the first product use period for participants randomized to Sequence B (i.e., participants who were randomized to receive FTC/TDF during their first product use period) or the second product use period for participants randomized to Sequence A (i.e., participants who were randomized to receive FTC/TDF during their second product use period).
Arm/Group | Dapivirine Vaginal Ring | FTC/TDF
Number analyzed (Participants) | 241 | 245
Participants
  Study Period 1 (Weeks 1-24): number analyzed (Participants) | 124 | 123
  Study Period 1 (Weeks 1-24): No grade 2+ AE | 36 | 36
  Study Period 1 (Weeks 1-24): At least one grade 2+ AE | 88 | 87
  Study Period 2 (Weeks 25-48): number analyzed (Participants) | 117 | 122
  Study Period 2 (Weeks 25-48): No grade 2+ AE | 22 | 28
  Study Period 2 (Weeks 25-48): At least one grade 2+ AE | 95 | 94
Statistical Analysis 1: Comparison: Dapivirine Vaginal Ring vs FTC/TDF; Comparison of the proportion of participants experiencing a grade 2 adverse event between products, with a null hypothesis of no difference; Test type: Superiority; p = 0.92, generalized estimating equation — the a priori threshold for statistical significance was <0.05; Poisson (log) link, adjusted for period, offset of number of visits per period, exchangeable correlation structure, and robust errors; incidence rate ratio = 1.01, 95% CI 2-sided [0.90 to 1.12] — The incidence rate ratio compares FTC/TDF to the dapivirine vaginal ring

2. Primary Outcome: Number of Participant-Visits With No Product Use
Description: During the study period where participants were randomized to use FTC/TDF they were assessed for FTC/TDF adherence by dried blood spot (DBS) at monthly visits. Results that were below the lower limit of detection (< 16.6 fmol/punch) were classified as no use of FTC/TDF during the preceding month, and detectable results (>= 16.6 fmol/punch) classified as at least some FTC/TDF use.
  During the study period where participants were randomized to use the dapivirine vaginal ring (VR) they were assessed for ring adherence by residual drug levels in returned VRs. Results that were less than or equal to a rate of 0.9mg dapivirine released per month were classified as no use of the VR during that month, and results greater than 0.9mg dapivirine release per month classified as at least some VR use.
Time Frame: Study periods 1 and 2
Population: Number of participant-visits during product use periods randomized to each product for which there is adherence data available.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Dapivirine Vaginal Ring | FTC/TDF
Number analyzed (Participants) | 241 | 245
Number analyzed (Visits) | 1407 | 1316
Visits
  Study Period 1: number analyzed (Participants) | 124 | 123
  Study Period 1: number analyzed (Visits) | 724 | 671
  Study Period 1: No use | 19 | 11
  Study Period 1: At least some use | 705 | 660
  Study Period 2: number analyzed (Participants) | 117 | 122
  Study Period 2: number analyzed (Visits) | 683 | 645
  Study Period 2: No use | 41 | 10
  Study Period 2: At least some use | 642 | 635

3. Secondary Outcome: Number of Participant-Visits Reporting Acceptability of Study Product
Description: During the study period where participants were randomized to use FTC/TDF they were asked to rate how much they liked using the tablets for HIV prevention (3 and 6 months after initiating the product).
  During the study period where participants were randomized to use the dapivirine vaginal ring they were asked to rate how much they liked using the ring for HIV prevention (3 and 6 months after initiating the product).
Time Frame: Study periods 1 and 2
Population: Number of participant-visits during product use periods randomized to each product for which there are responses to the question about acceptability.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Dapivirine Vaginal Ring | FTC/TDF
Number analyzed (Participants) | 241 | 245
Number analyzed (Visits) | 437 | 438
Visits
  Week 12: number analyzed (Participants) | 110 | 107
  Week 12: number analyzed (Visits) | 110 | 107
  Week 12: Like, or like very much | 105 | 72
  Week 12: Neither like nor dislike, dislike, or dislike very much | 5 | 35
  Week 24: number analyzed (Participants) | 111 | 105
  Week 24: number analyzed (Visits) | 111 | 105
  Week 24: Like, or like very much | 105 | 73
  Week 24: Neither like nor dislike, dislike, or dislike very much | 6 | 32
  Week 36: number analyzed (Participants) | 105 | 111
  Week 36: number analyzed (Visits) | 105 | 111
  Week 36: Like, or like very much | 91 | 93
  Week 36: Neither like nor dislike, dislike, or dislike very much | 14 | 18
  Week 48: number analyzed (Participants) | 111 | 115
  Week 48: number analyzed (Visits) | 111 | 115
  Week 48: Like, or like very much | 90 | 68
  Week 48: Neither like nor dislike, dislike, or dislike very much | 21 | 47

4. Secondary Outcome: Number of Participant-Visits With No Product Use
Description: During the study period where participants chose which product they used (i.e., Weeks 49-72) they were assessed for FTC/TDF adherence by dried blood spot (DBS) and/or dapivirine vaginal ring adherence by residual drug levels in returned VRs at monthly visits, depending on which product they chose. Results that were below the lower limit of detection (< 16.6 fmol/punch) were classified as no use of FTC/TDF during the preceding month, and detectable results (>= 16.6 fmol/punch) classified as at least some FTC/TDF use. Results that were less than or equal to a rate of 0.9mg dapivirine released per month were classified as no use of the VR during that month, and results greater than 0.9mg dapivirine release per month classified as at least some VR use.
Time Frame: Study period 3 (Weeks 49-72)
Population: Number of participant-visits during product choice period for which there is adherence data available.
Measure: Count of Units; unit: Visits
Units Other Than Participants: Visits
Arm/Group | Dapivirine Vaginal Ring | FTC/TDF
Number analyzed (Participants) | 164 | 87
Number analyzed (Visits) | 857 | 400
Visits
  No use | 57 | 19
  At least some use | 800 | 381

5. Secondary Outcome: Number of Participants Selecting Each Study Product
Description: During the third study product use period (i.e., Weeks 49-72) participants chose whether to use the dapivirine VR, FTC/TDF oral tablets, or neither product, and could change their decision throughout the 6 month period. Participants were categorized into one of four categories based on their selection pattern: always chose dapivirine VR, always chose FTC/TDF oral tablets, switched at least once (including switching to or from no product), and never chose either product.
Time Frame: Study period 3 (Weeks 49-72)
Population: All participants who attended at least one visit during study period 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: Dapivirine Vaginal Ring + FTC/TDF | Sequence B: FTC/TDF + Dapivirine Vaginal Ring
Number analyzed (Participants) | 120 | 118
Participants
  Always chose ring | 66 | 71
  Always chose tablets | 35 | 27
  At least one switch | 17 | 13
  Never chose ring or tablets | 2 | 7

6. Secondary Outcome: Percentage of Participants Reporting Preference for Dapivirine VR as Compared to FTC/TDF Oral Tablets
Description: Participants were asked "would you prefer to use the ring or the tablets for HIV prevention?" at their enrollment, Month 12, and product use end visit (Month 18) visits.
Time Frame: All three study periods (enrollment, month 12, and month 18 study visits)
Population: The analysis population is all participants who completed the questionnaire at the visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequence A: Dapivirine Vaginal Ring + FTC/TDF | Sequence B: FTC/TDF + Dapivirine Vaginal Ring
Number analyzed (Participants) | 124 | 123
Participants
  Enrollment: Preferred ring | 51 | 43
  Enrollment: Preferred tablets | 43 | 57
  Enrollment: Either product equally | 29 | 18
  Enrollment: Neither product | 0 | 4
  Enrollment: Skipped question | 1 | 1
  Month 12: number analyzed (Participants) | 116 | 111
  Month 12: Preferred ring | 74 | 76
  Month 12: Preferred tablets | 37 | 30
  Month 12: Either product equally | 5 | 2
  Month 12: Neither product | 0 | 2
  Month 12: Skipped question | 0 | 1
  Month 18: number analyzed (Participants) | 115 | 108
  Month 18: Preferred ring | 67 | 66
  Month 18: Preferred tablets | 35 | 33
  Month 18: Either product equally | 13 | 5
  Month 18: Neither product | 0 | 4
  Month 18: Skipped question | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the duration of participants' time on study (18 months)
Description: The "Any Event in SOC" rows summarize the total number of adverse events within an SOC. These events are also summarized using the specific Adverse Event Term for the event.
Groups:
- Dapivirine Vaginal Ring (Periods 1 and 2): The period during the first two product use periods where the participant was randomized to use the dapivirine ring. This is the first product use period for participants randomized to Sequence A (i.e., participants who were randomized to receive the dapivirine vaginal ring during their first product use period) or the second product use period for participants randomized to Sequence B (i.e., participants who were randomized to receive the dapivirine vaginal ring during their second product use period).
- FTC/TDF (Periods 1 and 2): The period during the first two product use periods where the participant was randomized to use FTC/TDF. This is the first product use period for participants randomized to Sequence B (i.e., participants who were randomized to receive FTC/TDF during their first product use period) or the second product use period for participants randomized to Sequence A (i.e., participants who were randomized to receive FTC/TDF during their second product use period).
- Choice Period (Period 3): The third study period was intended to assess product choice and not inform the safety profile of the products. As such, the third study period was designed to allow participants to choose the dapivirine ring, oral FTC/TDF, or neither product. Because participants could also choose to switch between these three options throughout the study period without any washout period between switches, it is not possible to ascribe AEs to a specific product. Therefore, adverse events occurring during this period are combined.
Arm/Group | Dapivirine Vaginal Ring (Periods 1 and 2) | FTC/TDF (Periods 1 and 2) | Choice Period (Period 3)
All-Cause Mortality (participants affected / at risk) | 0/241 | 0/245 | 0/238
Serious Adverse Events (participants affected / at risk) | 0/241 | 3/245 | 3/238
Other Adverse Events (participants affected / at risk) | 205/241 | 219/245 | 203/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Vaginal Ring (Periods 1 and 2) (N=241) | FTC/TDF (Periods 1 and 2) (N=245) | Choice Period (Period 3) (N=238)
Any Event in SOC (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapivirine Vaginal Ring (Periods 1 and 2) (N=241) | FTC/TDF (Periods 1 and 2) (N=245) | Choice Period (Period 3) (N=238)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 4 (4) | 2 (2)
Anaemia of pregnancy (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Any Event in SOC (Blood and lymphatic system disorders) | 6 (7) | 7 (7) | 5 (6)
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Swelling of eyelid (Eye disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 16 (16) | 30 (33) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Any Event in SOC (Gastrointestinal disorders) | 38 (46) | 104 (189) | 29 (39)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 29 (34) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (12) | 59 (74) | 9 (10)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 31 (37) | 10 (10)
Any Event in SOC (General disorders) | 6 (6) | 17 (18) | 4 (4)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 2 (2) | 12 (13) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 1 (1)
Implant site pain (General disorders) | 1 (1) | 1 (1) | 0 (0)
Implant site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 0 (0)
Suprapubic pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Acute HIV infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Any Event in SOC (Infections and infestations) | 141 (271) | 130 (257) | 150 (262)
Bacterial vaginosis (Infections and infestations) | 15 (15) | 12 (13) | 11 (11)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 7 (7)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Cervicitis (Infections and infestations) | 2 (2) | 1 (1) | 4 (4)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Dermatophytosis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Fungal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 3 (4)
Gastroenteritis (Infections and infestations) | 8 (8) | 8 (9) | 7 (7)
Genitourinary chlamydia infection (Infections and infestations) | 61 (71) | 58 (67) | 63 (82)
Genitourinary tract gonococcal infection (Infections and infestations) | 26 (27) | 31 (36) | 29 (33)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 3 (3) | 5 (5)
Malaria (Infections and infestations) | 8 (10) | 12 (17) | 8 (8)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pelvic inflammatory disease (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 5 (5)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Skin candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 2 (2) | 4 (4) | 3 (4)
Syphilis (Infections and infestations) | 3 (3) | 4 (4) | 4 (4)
Tinea faciei (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tonsillitis (Infections and infestations) | 5 (5) | 2 (2) | 0 (0)
Trichomoniasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Typhoid fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 29 (30) | 16 (18) | 12 (12)
Upper respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 23 (27) | 19 (20) | 22 (22)
Varicella (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulval abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 20 (22) | 13 (14) | 12 (13)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Vulvovaginitis trichomonal (Infections and infestations) | 25 (27) | 22 (28) | 19 (22)
Any Event in SOC (Injury, poisoning and procedural complications) | 3 (3) | 8 (8) | 8 (8)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Burns first degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ear injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Human bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Any Event in SOC (Investigations) | 78 (95) | 90 (109) | 89 (102)
Blood creatinine increased (Investigations) | 9 (9) | 12 (13) | 14 (14)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 5 (5) | 3 (3) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 73 (75) | 83 (85) | 76 (76)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 2 (3)
Neutrophil count decreased (Investigations) | 3 (3) | 3 (3) | 6 (6)
Platelet count decreased (Investigations) | 1 (1) | 2 (3) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Metabolism and nutrition disorders) | 6 (6) | 12 (14) | 6 (6)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 9 (10) | 6 (6)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 6 (6) | 12 (12) | 7 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 5 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 3 (3)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 2 (2)
Any Event in SOC (Nervous system disorders) | 38 (47) | 87 (119) | 23 (26)
Dizziness (Nervous system disorders) | 9 (9) | 47 (48) | 5 (5)
Headache (Nervous system disorders) | 28 (31) | 56 (67) | 17 (18)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 6 (6) | 2 (3) | 3 (3)
Any Event in SOC (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
Haemorrhage in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
Adjustment disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Any Event in SOC (Renal and urinary disorders) | 5 (5) | 6 (7) | 4 (4)
Dysuria (Renal and urinary disorders) | 3 (3) | 6 (6) | 3 (3)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Post micturition dribble (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Any Event in SOC (Reproductive system and breast disorders) | 70 (107) | 40 (56) | 46 (60)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cervical discharge (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 7 (7) | 5 (5) | 11 (11)
Dyspareunia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Genital discomfort (Reproductive system and breast disorders) | 2 (2) | 2 (2) | 0 (0)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Genital ulceration (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 3 (3) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 8 (11) | 1 (1) | 1 (1)
Nipple pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 4 (4) | 4 (4) | 2 (2)
Perineal rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Premenstrual headache (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 31 (33) | 20 (22) | 22 (25)
Vaginal lesion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal odour (Reproductive system and breast disorders) | 22 (22) | 5 (5) | 3 (3)
Vaginal polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulval disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulval ulceration (Reproductive system and breast disorders) | 3 (3) | 3 (3) | 1 (1)
Vulvar erosion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 4 (4) | 0 (0) | 4 (4)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 9 (10) | 3 (3) | 7 (7)
Vulvovaginal rash (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (6) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 11 (11) | 14 (14) | 9 (11)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (2)
Any Event in SOC (Social circumstances) | 1 (1) | 3 (3) | 1 (1)
Victim of sexual abuse (Social circumstances) | 1 (1) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/55/NCT03593655/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/55/NCT03593655/SAP_001.pdf